CLINICAL TRIAL: NCT02935660
Title: A Prospective, Multi-Center Pivotal Clinical Evaluation of a Novel Multi-Wavelength Laser for Tattoo Removal
Brief Title: Multi-Wavelength Laser Tattoo Removal Pivotal Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cutera Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-16-EN13
Record Dates: First submitted 2016-10-14; First posted 2016-10-17 (Estimated); Results first posted 2023-09-26 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Tattoo Removal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Treatment with investigational Cutera enlighten laser for tattoo removal
  Interventions: Device: enLighten Laser

INTERVENTIONS:
Device: enLighten Laser — Laser tattoo removal treatment

SUMMARY:
Multi-center study to evaluate the safety and efficacy of an investigational version of the Cutera enlighten laser that offers multiple wavelengths for tattoo removal

DETAILED DESCRIPTION:
A multi-center prospective, open-label, uncontrolled pivotal study to evaluate the safety and efficacy of an investigational version of the Cutera enlighten laser that offers multiple wavelengths for tattoo removal.

ELIGIBILITY:
Inclusion Criteria:

* Female or Male, 18 to 65 years of age (inclusive).
* Fitzpatrick Skin Type I - VI.
* Target tattoo contains single or multi-color ink, and must include blue and/or green ink.
* Target tattoos must be older than 1 year.
* Target treatment area not to exceed 12 square inches.
* Subject must be able to read, understand and sign the Informed Consent Form.
* Must be willing and able to adhere to the treatment and follow-up schedule and post-treatment care instructions.
* Wiling to cover tattoos with a bandage or clothing; and/or have very limited sun exposure and use an approved sunscreen of SPF 50 or higher on the treated area starting 2 to 4 weeks before the treatment and/or every day for the duration of the study, including the follow-up period.
* Willing to have digital photographs taken of the treatment area and agree to use of photographs for presentation, educational or marketing purposes.
* Agree to not undergo any other procedure(s) for tattoo removal during the study (as applicable).
* Post-menopausal or surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment and during the entire course of the study, and no plans to become pregnant for the duration of the study.

Exclusion Criteria:

* Participation in a clinical trial of a drug or another device in the target area during the study.
* Target tattoo contains only black ink.
* History of allergic reaction to pigments following tattooing.
* History of allergy to local anesthetics.
* History of allergy to topical antibiotics.
* History of malignant tumors in the target area.
* Skin abnormalities in the target area, e.g., cuts, scrapes, wounds, scars, large moles.
* Pregnant and/or breastfeeding.
* Having an infection, dermatitis or a rash in the treatment area.
* Significant concurrent illness, such as diabetes mellitus or cardiovascular disease, e.g., uncontrolled hypertension.
* Suffering from coagulation disorders or taking prescription anticoagulation medications.
* History of keloid scarring, hypertrophic scarring or of abnormal wound healing.
* History of immunosuppression/immune deficiency disorders or currently using immunosuppressive medications per investigator's discretion.
* History of vitiligo, eczema, or psoriasis.
* History of connective tissue disease, such as systemic lupus erythematosus or scleroderma.
* History of seizure disorders due to light.
* Any use of medication that is known to increase sensitivity to light according to Investigator's discretion.
* History of disease stimulated by heat, such as recurrent herpes simplex and/or herpes zoster (shingles) in the treatment area, unless treatment is conducted following a prophylactic regimen.
* History of radiation to the treatment area or undergoing systemic chemotherapy for the treatment of cancer.
* History of pigmentary disorders, particularly tendency for hyper- or hypo-pigmentation.
* Systemic use of corticosteroid or isotretinoin, as applicable, within 6 months of study participation.
* Anytime in life, having used gold therapy (gold salts) for disorders such as rheumatologic disease or lupus.
* Excessively tanned in areas to be treated or unable/unlikely to refrain from tanning during the study.
* Current smoker or history of smoking within 6 months of study participation.
* As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Cutera Research Clinic, Brisbane, California
  - Skin Care Physicians, Chestnut Hill, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment
Started | 27
Completed | 25
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 27
Age, Continuous [Mean (Full Range); unit: years] | 38.7 [24 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 1
  White | 21
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Tattoo Clearing as Rated by Blinded Evaluator
Description: Percentage of subjects with tattoo ink clearing of at least 50% or more at 6 weeks post-final treatment
Time Frame: 6 weeks post-final treatment, approximately 7 months after study start
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 25
Participants | 21

2. Secondary Outcome: Degree of Overall Tattoo Ink Clearing at 6 Weeks Post-final Treatment as Assessed by the Investigator (Physician's Global Assessment of Improvement).
Description: Physician's Global Assessment of Improvement (min=0; max=4) Higher scores mean better outcomes
Time Frame: 6 weeks post-final treatment, approximately 7 months after study start
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 25
score on a scale | 3.43 (0.7)

3. Secondary Outcome: Subject Satisfaction Levels at 6 Weeks Post-final Treatment
Time Frame: 6 weeks post-final treatment, approximately 7 months after study start
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 13
Participants
  number of subjects reporting they were "extremely satisfied" or "satisfied" with level of clearing | 9
  number of subjects reporting they were neutral with level of clearing | 4
  number of subjects who said they would the investigational treatment again | 11

4. Secondary Outcome: Subject Pain During Treatment
Description: Numeric Pain Rating Scale (Min=0; Max=10) Higher scores indicate worse outcomes Pain values from all treatment visits and subjects were combined and averaged.
Time Frame: Reported by subject at the end of each treatment visit, up to 5 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 27
score on a scale | 4.2 (2.9)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected 6 weeks post final laser treatment, up to an average of 7 months
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 27/27
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=27)
Erythema (Skin and subcutaneous tissue disorders) | 27
Edema (Skin and subcutaneous tissue disorders) | 27
Frosting (Skin and subcutaneous tissue disorders) | 27
Crusting (Skin and subcutaneous tissue disorders) | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-02): https://cdn.clinicaltrials.gov/large-docs/60/NCT02935660/Prot_SAP_000.pdf